CLINICAL TRIAL: NCT03304431
Title: Evaluation of the Effect of 10% Lidocaine Spray on Hemodynamic Response and EKG Parameter Performed Before Endotracheal Intubation in Patients Undergoing Coronary Artery Bypass Graft Operation
Brief Title: Evaluation of the Effect of 10% Lidocaine Spray Undergoing Coronary Artery Bypass Graft Operation
Acronym: ELCABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AbantIBU mb5
Record Dates: First submitted 2017-08-07; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Diseases; Lidocaine Causing Adverse Effects in Therapeutic Use; Tracheal Intubation Morbidity
Keywords: QT dispersion; topical lidocaine; P-wave values
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The induction of group L will be performed 5 minutes after administration of 10% topical lidocaine (Vemcaine pump spray 10% 50 ml) 160 mg (16 puffs).
Who Masked: Outcomes Assessor
Masking Description: QTc (corrected QT), QT dispersion (QTd), P wave dispersion will calculated by a blind researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group(Group C) (No Intervention): After pre-oxygenation, anesthesia induction will be performed with intravenous administration of 2 μg / kg fentanyl, 2 mg/kg propofol, 0.6 mg/kg rocuronium bromide (Esmeron 5 mg vial, Organon Oss Holanda).
- Group L (Other): The induction of group L will be performed 5 minutes after administration of 10% topical lidocaine (Lidocaine pump spray 10% 50 ml) 160 mg (16 puffs) application
  Interventions: Drug: Orotracheal Lidocaine Oral Spray application

INTERVENTIONS:
Drug: Orotracheal Lidocaine Oral Spray application — The induction of group L will be performed 5 minutes after administration of 10% topical lidocaine (Lidocaine pump spray 10% 50 ml) 160 mg (16 puffs) application
  Arms: Group L

SUMMARY:
In patients undergoing coronary bypass surgery; 10% topical lidocaine administered endotracheally before intubation is to investigate the effect of hemodynamic response and EKG paramater after intubation.

DETAILED DESCRIPTION:
This prospective randomized double-blind study consisted of 60 volunteers undergoing coronary artery bypass surgery. Patients will be randomized and divided into two groups as control (Group C) = 30) and topical lidocaine group (Group L) = 30). Two intravenous 18-gauge (G) cannula will be inserted to all patients. Premedication will be provided with 0.03 mg/kg intravenous (iv) midazolam (Dormicum 1 mg/ml, Roche preparations Inc., Istanbul Turkey) and 50 mcg fentanyl and patients will be given 2 L / min O2 via nasal cannula. Radial artery cannulation will be performed by applying an Allen Test with 20G cannula under topical anesthesia. heart rate (HR), mean arterial pressure (MAB), peripheral oxygen saturation (SpO2) will be recorded. Induction of group C will be performed after preoperative preparation. No intervention will be made in group c and standard anesthesia protocol will be applied.

Group L (intervention group) Oral-tracheal lidocaine spray will be applied. The induction of group L will be performed 5 minutes after administration of 10% topical lidocaine (Lidocaine pump spray 10% 50 ml) 160 mg (16 puffs) . After pre-oxygenation, anesthesia induction will be performed with intravenous administration of 2 μg / kg fentanyl, 2 mg/kg propofol, 0.6 mg/kg rocuronium bromide (Esmeron 5 mg vial, Organon Oss Holanda). Tracheal intubation of all patients will be performed by an experienced anesthesiologist after providing adequate relaxation. Anesthesia will be maintained with sevoflurane(Forane, Abbott, İstanbul Türkiye) % 2 in a 50% Air +50% O2 mixture. ECG recording of participants will be performed before (baseline) and after one minute from induction and at the first and third minutes following intubation. Hemodynamic measurements and record (MAB, HR, SpO2) will be performed at baseline one minute after the induction of anesthesia as well as at 1,3,5,10 min after tracheal intubation. Before the ECG analysis, all participants will be blinded by closing their group names on the ECG recording. QTc (corrected QT,), QT intarvale dispersion (QTd), P wave dispersion will calculated by a blind researcher within a 12-lead ECG recording (velocity: 25 mm / sec, Amplitude: 10 mm / mV). QTd , was the difference between the longest QT intervale(QT max.) durations and shortest QT intervale(QT min.) durations(msec); P wave dispersion, was the difference between the longest and shortest P-wave durations(msec); QTc interval was calculated using Bazett's formula (QTc = QT/√RR).)

ELIGIBILITY:
Inclusion Criteria:

* 50-75 between age patients
* ASA status III patients
* patients undergoing coronary artery bypass graft operation

Exclusion Criteria:

* cardiomyopathy,
* arrhythmia,
* valvular disease,
* electrolyte disorders
* chronic liver and kidney diseases
* use of medication that led to extended QT intervals

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
ECG parameter | baseline, one minute from induction,first and third minutes following intubation
  P wave dispersion was the difference between the longest and shortest P-wave durations (msec); )

SECONDARY OUTCOMES:
hemodynamic response | baseline, after anesthesia induction one minute, after tracheal intubation 1 minute, 3 minute, 5 minute, 10 minute
  heart rate (beats / minute)
hemodynamic response | baseline, after anesthesia induction one minute, after tracheal intubation 1 minute,3 minute, 5 minute, 10 minute
  mean arterial pressure(mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: murat bilgi, Principal Investigator — Abant Izzet Baysal University Medical School, Bolu, TURKEY
Locations (1):
- Abant Izzet Baysal University Medical School,, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hanci V, Yurtlu S, Karabag T, Okyay D, Hakimoglu S, Kayhan G, Buyukuysal C, Ayoglu H, Ozkocak Turan I. Effects of esmolol, lidocaine and fentanyl on P wave dispersion, QT, QTc intervals and hemodynamic responses to endotracheal intubation during propofol induction: a comparative study. Braz J Anesthesiol. 2013 May-Jun;63(3):235-44. doi: 10.1016/S0034-7094(13)70223-X. English, Portuguese, Spanish. PMID 23683444
- [Derived] Bilgi M, Velioglu Y, Yoldas H, Cosgun M, Yuksel A, Karagoz I, Yildiz I, Es A, Caliskan D, Erdem K, Demirhan A. Effects of Lidocaine Oropharyngeal Spray Applied Before Endotracheal Intubation on QT Dispersion in Patients Undergoing Coronary Artery Bypass Grafting: A Prospective Randomized Controlled Study. Braz J Cardiovasc Surg. 2020 Jun 1;35(3):291-298. doi: 10.21470/1678-9741-2019-0112. PMID 32549100
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/?term=Effects+of+esmolol%2C+lidocaine+and+fentanyl+on+P+wave+dispersion%2C+QT%2C+QTc+intervals+and+hemodynamic+responses+to+endotracheal+intubation+during+propofol+induction%3A+a+comparative+study